CLINICAL TRIAL: NCT02437929
Title: Procedural Pain in Palliative Care: Prevalence, Intensity and Treatment. A Prospective, Cross-sectional, Multicenter, National Study
Brief Title: Procedural Pain in Palliative Care: Prevalence, Intensity and Treatment
Status: Completed | Type: Observational
Sponsor: Antea Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PCPP02
Record Dates: First submitted 2015-04-30; First posted 2015-05-08 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2015-12

CONDITIONS: Breakthrough Pain; Pain Due to Certain Specified Procedures; Pain; Cancer; Terminal Disease
MeSH Terms: conditions — Breakthrough Pain; Pain; Neoplasms | interventions — Patient Positioning; Urinary Catheterization

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving standard procedures
  Interventions: Procedure: Mobilization; Procedure: Positioning; Procedure: Personal Hygiene Care; Procedure: Bladder catheterization; Procedure: Wound care; Procedure: Subcutaneous drugs administration

INTERVENTIONS:
Procedure: Mobilization
Procedure: Positioning
Procedure: Personal Hygiene Care
Procedure: Bladder catheterization
Procedure: Wound care
Procedure: Subcutaneous drugs administration

SUMMARY:
This study aims to assess self reported procedural pain compared with background pain and evaluate pain intensity differences across six standard procedures. Besides, rescue and preventive treatments used to control procedural pain will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving the procedures included in this study as a part of their standard care
* Patients that have expressed their consent to participate to the study by signing the informed consent document

Exclusion Criteria:

* Very serious or unstable clinical conditions with a Karnofsky Performance Status Index (KPS) < 20
* Presence of neurological or psychiatric conditions, due to the original disease or concomitant diseases, interfering with the patient's level of consciousness or with judgment, such as to compromise compliance with the study protocol;
* Not adequately controlled background pain (average NRS in the last 24 hours is > 4)
* Emergency procedures or procedures performed during night time (from 8 p.m. until 8 a.m)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Terminally ill patients, cancer and non-cancer, admitted in a palliative care service (inpatients or outpatients), that are undergoing at least one procedure considered in the study, as a part of their Individual Care Plan (ICP).
Sampling Method: Non-Probability Sample
Enrollment: 1079 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
11 Points - Numerical Rating Scale (NRS); change in baseline pain intensity during the procedure (of 3 points NRS or higher) | Participants will be followed 10 minutes before the procedure, for the duration of the procedure and ten minutes after, an expected average of 1 hour
  Self reported pain intensity 10 minutes before the procedure, during the procedure (measured immediately after that the procedure is performed), 10 minutes after the procedure. Each item is scored 0-10 (0 = no pain; 10 = worst possible pain).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Casale, Medicine, Principal Investigator — Antea Foundation
Locations (1):
- San Marco hospice, Latina, Italy

IPD SHARING:
Plan to Share IPD: No